CLINICAL TRIAL: NCT05278754
Title: Independent Predictors Analysis and Model Construction of Cavitary Central Lung Cancer: a Retrospective, Multicenter Trial
Brief Title: Independent Predictors Analysis and Model Construction of Cavitary Central Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Central Hospital of Lishui City (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other); The Second Affiliated Hospital of Medical College of Zhejiang University (Unknown); Affiliated Hospital of Xinjiang Medical University (Unknown)
Responsible Party: Sponsor
Other Study IDs: ZJLS-KLDMIR-22004
Record Dates: First submitted 2022-02-10; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Central Lung Cancer
Keywords: Central Lung Cancer; Cavity; Predictor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a retrospective, multicenter clinical study. The main goal is to identify the risk factors for cavity formation in central-type lung cancer lesions, and to construct a prediction model for cavity formation in central-type lung cancer lesions based on the above risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Age：older than 18 years；
2. Clinical or pathologically confirmed central lung cancer;
3. Lesions without cavities at first diagnosis of central lung cancer;
4. Performed complete laboratory and imaging research at the first diagnosis of the central lung cancer;
5. Patients with cavities formation during follow up, and the cavities were independently confirmed by at least 3 imaging experts;
6. Patients with complete medical records;

Exclusion Criteria:

1. Patients suffering other malignant tumors;
2. Patients missing the imaging data;
3. Patients missing the clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter study. Patients from Lishui Central Hospital of Zhejiang Province, the Second Affiliated Hospital of Medical College of Zhejiang University, and Affiliated Hospital of Xinjiang Medical University who meet the above criteria will be included in this study
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-03-12 (Estimated); Primary Completion 2022-05-12 (Estimated); Study Completion 2022-08-12 (Estimated)

PRIMARY OUTCOMES:
Formation of cavities in the central lung cancer, assessed up to 18 months. | Time from enrollment to the time of cavities formation, assessed up to 18 months.
  Time from enrollment to the time of cavities formation, assessed up to 18 months.

SECONDARY OUTCOMES:
Hemoptysis in patients with central lung cancer, assessed up to 18 months. | Time from enrollment to hemoptysis, assessed up to 18 months.
  Time from enrollment to hemoptysis, assessed up to 18 months.

IPD SHARING:
Plan to Share IPD: Yes
Statistical analysis plan, informed consent form, and clinical study report can be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within six months after the trial is completed.
Access Criteria: Shared data is not available for downloading, but can only be browsed. To download the data, you must contact the researchers. Shared data does not provide any private information of the participants.